CLINICAL TRIAL: NCT00364247
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Multiple Doses of CG5503 Immediate-Release Formulation in the Treatment of Acute Pain From Bunionectomy Followed by a Voluntary Open-Label Extension
Brief Title: A Study to Evaluate the Effectiveness and Safety of Tapentadol(CG5503) in the Treatment of Acute Pain From Bunionectomy Compared With Placebo Followed by a Voluntary Open Label Extension for Safety.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR011215
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Arthralgia; Bunion; Hallux Valgus; Pain Assessment; Tapentadol
Keywords: Acute pain; bunionectomy
MeSH Terms: conditions — Arthralgia; Bunion; Hallux Valgus; Acute Pain

INTERVENTIONS:
Drug: CG5503 IR;tapentadol

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of the administration of 3 different dose levels of CG5503 compared with oxycodone and with placebo in patients who have had a bunionectomy, and to assess the safety of the drug for 9 days after patients are discharged from the hospital.

DETAILED DESCRIPTION:
Patients undergoing bunionectomy often experience moderate to severe acute pain post-surgery. Normally such pain is controlled when patients receive repeated doses of opioid analgesics. However, opioid therapy is commonly associated with side effects such as nausea, vomiting, sedation, constipation, addiction, tolerance, and respiratory depression. CG5503, a newly synthesized drug also acts as a centrally acting analgesic but has a dual mode of action. The aim of this study is to investigate the effectiveness (level of pain control) and safety (side effects) of 3 dose levels of CG5503 Immediate Release (IR) compared to no drug (placebo) or one dose level of oxycodone (an opioid commonly used to treat post-surgical pain). This study is a randomized (patients are assigned different treatments based on chance), double-blind (neither investigator nor patient will know which treatment is received), active- and placebo-controlled, parallel-group, multicenter study to evaluate treatment of the acute pain from bunionectomy. The study will include a blinded 72 hour inpatient phase immediately following bunionectomy, during which patients will be treated with either 50-, 75-, or 100-mg CG5503 IR base, a placebo, or 15-mg oxycodone IR, and pain intensity and pain relief will be periodically assessed. Following this phase, patients wishing to continue treatment with CG5503 IR may enter an outpatient voluntary nonrandomized, open-label extension phase for 9 days when they will receive 50- or 100-mg CG5503 IR. Assessments of pain relief include the pain intensity numeric rating scale (PI), pain relief numeric rating scale (PAR), and patient global impression of change scale (PGIC). Safety evaluations include monitoring of adverse events, physical examinations, and clinical laboratory tests. Venous blood samples will be collected for the determination of serum concentrations of CG5503 and oxycodone. The null hypothesis for the study is that efficacy results for all CG5503 IR dosage groups are equal to placebo based on the mean sum of pain intensity difference at 48 hours. The alternative study hypothesis is that at least 1 dose strength of CG5503 will be different from placebo in controlling pain at 48 hours. CG5503 IR 50, or 75, or 100 mg (of the base), or oxycodone 15 mg, or placebo: 1 capsule taken every 4 to 6 hours during the 72-hour postsurgery phase of the study; and CG5503, 50 mg capsules, 1 to 2 tablets taken by mouth every 4 to 6 hours for up to 9 days during the open label portion of the study. All doses of study treatment will be taken with approximately 120 mL of water with or without food.

ELIGIBILITY:
Inclusion Criteria:

* Patients must undergo primary unilateral first metatarsal bunionectomy
* pain intensity must be moderate to severe following stoppage of a continuous popliteal sciatic block (a nerve block with local anesthetic that numbs the foot)
* female patients must be postmenopausal, surgically sterile, or practicing an effective method of birth control if they are sexually active.

Exclusion Criteria:

* Patients will be excluded from the study if they have a history of seizure disorder or epilepsy
* history of malignancy within the past 2 years before starting the study
* history of alcohol or drug abuse
* evidence of active infections that may spread to other areas of the body
* clinical laboratory values reflecting moderate or severe renal insufficiency
* currently treated with anticonvulsants, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), neuroleptics, or serotonin norepinephrine reuptake inhibitor (SNRI).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness outcome for this study is SPID48 (i.e., the sum of pain intensity difference at 48 hours relative to the first dose).

SECONDARY OUTCOMES:
Secondary effectiveness outcomes include, among others, the effect of CG5503 IR on the time to the need for the first rescue pain medication during the double-blind treatment period, and the SPID at 12, 24, and 72 hours relative to first dose.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Daniels SE, Upmalis D, Okamoto A, Lange C, Haeussler J. A randomized, double-blind, phase III study comparing multiple doses of tapentadol IR, oxycodone IR, and placebo for postoperative (bunionectomy) pain. Curr Med Res Opin. 2009 Mar;25(3):765-76. doi: 10.1185/03007990902728183. PMID 19203298
- See also: A Study to Evaluate the Effectiveness and Safety of Tapentadol(CG5503) in the Treatment of Acute Pain From Bunionectomy Compared With Placebo Followed by a Voluntary Open Label Extension for Safety. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=727&filename=CR011215_CSR.pdf